CLINICAL TRIAL: NCT06852014
Title: Effects of Peptamen 1.6 in Malnourished Patients (or in Risk) With Pancreatic Neoplasia Undergoing Cephalic Pancreaticoduodenectomy (CPD): A Study Mechanistic.
Brief Title: Effects of Peptamen 1.6 in Malnourished Patients (or at Risk) With Pancreatic Neoplasia Undergoing Cephalic Pancreaticoduodenectomy (CPD): A Mechanistic Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PEP-NUTRIDPC trial
Record Dates: First submitted 2025-02-13; First posted 2025-02-28 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Pancreatic Cancer, Adult; Cephalic Duodenopancreatectomy
Keywords: Pancreatic cancer; malnutrition; pancreaticoduodenectomy; oral nutritional supplement; gut microbiota; organoids
MeSH Terms: conditions — Pancreatic cancer, adult; Pancreatic Neoplasms; Malnutrition

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in a 1:1 ratio
Who Masked: Participant, Investigator
Masking Description: Patients will take Peptamen 1,6 and Resource HP/HC de forma secuencial pero con un orden predeterminado as assigned at randomization . For this purpose, identical formats will be used and neither the participant nor the researcher will know their content.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EXPERIMENTAL GROUP A (Nutritional supplement order A --> B) (Experimental)
  Interventions: Dietary Supplement: Dietary Supplement: Experimental Treatment with nutritional suplement A + nutritional suplement B
- EXPERIMENTAL : EXPERIMENTAL GROUP B (Nutritional supplement order B --> A) (Experimental)
  Interventions: Dietary Supplement: Dietary Supplement: Dietary Supplement: Experimental Treatment with nutritional suplement B + nutritional suplement A

INTERVENTIONS:
Dietary Supplement: Dietary Supplement: Experimental Treatment with nutritional suplement A + nutritional suplement B — Intervention group will receive a nutritional formula A and, after 1-week washout period, will receive a nutritional formula B
  Arms: EXPERIMENTAL GROUP A (Nutritional supplement order A --> B)
Dietary Supplement: Dietary Supplement: Dietary Supplement: Experimental Treatment with nutritional suplement B + nutritional suplement A — Intervention group will receive a nutritional formula B and, after 1-week washout period, will receive a nutritional formula A
  Arms: EXPERIMENTAL : EXPERIMENTAL GROUP B (Nutritional supplement order B --> A)

SUMMARY:
Malnutrition is a common challenge in patients with pancreatic cancer undergoing cephalic pancreaticoduodenectomy (CPD), impacting postoperative recovery and overall prognosis. Nutritional support plays a crucial role in optimising metabolic, inflammatory, and digestive outcomes. This randomised, double-blind, crossover clinical trial aims to evaluate the effects of Peptamen 1.6, a hydrolysed whey protein-based enteral formula, compared to Resource HP/HC, a high-protein and high-calorie polymeric formula, in malnourished or at-risk patients with pancreatic cancer undergoing PD.

The study comprises both in vivo and in vitro analyses. The in vivo component will assess the impact of Peptamen 1.6 on digestive tolerance, amino acid absorption, nutritional status, metabolic profile, inflammatory markers, and gut microbiota composition. The in vitro component will utilise human intestinal organoid models to explore how enteral nutrition formulations influence intestinal permeability and metabolism, with a focus on microbiota interactions.

Primary outcomes include improvements in metabolic status, assessed through serum biomarkers (albumin, immune markers, intestinal permeability, and myosin profile), inflammatory status via peripheral blood mononuclear cells (PBMCs), and microbiota shifts in faecal samples. Additionally, adherence to treatment, digestive tolerance, and changes in body composition will be monitored using bioelectrical impedance, dynamometry, and functional mobility tests.

By elucidating the mechanisms through which different enteral nutrition strategies influence clinical, physiological, and molecular parameters, this study aims to enhance personalised nutritional interventions for patients with pancreatic cancer. The findings could contribute to optimising nutritional support strategies, ultimately improving patient outcomes following CPD.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory patients who are malnourished or at risk of malnutrition, with a confirmed diagnosis of neoplasms of the periampullary region, pancreas, and duodenum, or pancreatic cancer, and who have undergone cephalic pancreaticoduodenectomy (CPD).
* No prior neoadjuvant treatment (preoperative chemotherapy or radiotherapy): Patients must not have received neoadjuvant therapy as these treatments can affect metabolism, nutritional status, and gut microbiota, potentially interfering with the objectives of the study's nutritional intervention.

Exclusion Criteria:

* Refusal to sign informed consent: Informed consent is a mandatory requirement for study participation. Any patient unwilling to participate voluntarily will be excluded.
* Patients who underwent surgery more than three months ago will be excluded, as the nutritional intervention must begin in the immediate postoperative period to adequately evaluate its impact on nutritional and metabolic status.
* Presence of severe cardiac disease, nephropathy, or other severe comorbidities: Conditions such as severe cardiac disease, renal failure, or comorbidities that could induce malnutrition or impair the patient's ability to tolerate nutritional treatment will be exclusion criteria. These conditions may interfere with assessing the effects of nutritional supplementation in the context of pancreatic cancer treatment.
* Diarrhoea associated with antibiotics, laxatives, or osmotically active agents: Diarrhoea caused by medications may alter nutrient absorption and affect tolerance to the nutritional supplement, potentially skewing results attributable solely to the nutritional intervention.
* Treatment with other nutritional support: Patients receiving other oral nutritional supplement, enteral or parenteral nutrition will be excluded, as interactions with the studied formula could confound the efficacy results of the study's nutritional intervention.
* Pregnancy or possibility of becoming pregnant.
* Type 1 or Type 2 diabetes with HbA1c >8%.
* Galactosaemia, fructosaemia, or allergies to components of the nutritional supplement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-29 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Adherence to nutritional treatment | At weeks 6 and 13
  Categorized based on the average daily consumption compared to the prescribed volume (200 ml per bottle):
  * Full content (200 ml/bottle)
  * 2/3 content (150 ml/bottle)
  * 1/2 content (100 ml/bottle)
  * 1/4 content (50 ml/bottle)
  Patients will self-report their average daily consumption (ml/day).
Natural food intake | At weeks 6 and 13
  Patients will report their food intake over the previous week, categorized into quartiles (%) relative to:
  * Pre-illness consumption
  * Perceived normal intake for patients without supplementation
    * ALL -100%
    * 3/4 - 75%
    * HALF - 50%
    * ¼ - 25%
    * NONE - 0%
Tolerance to nutritional treatment | At weeks 6 and 13
  Evaluated based on the frequency of gastrointestinal symptoms (e.g., nausea, vomiting, reflux, abdominal pain, flatulence, satiety, constipation, and stomach heaviness) within two hours of supplement consumption.
  Symptoms classified as:
  * Never
  * Rarely
  * Sometimes
  * Frequently
  * Always
  Bivariate analysis will classify tolerance as:
  * Good (no symptoms)
  * Poor (presence of any gastrointestinal symptoms)
Change in aminoacids: Ala, Glu, Asp, Pro, Phe, Leu/Ile, Val, Tyr, Met, Cit, Arg, Gly, and Orn | At baseline and in weeks 6, 7, and 13
  Aminoacids measured in µmol/L
Change in IL-6 and TNF-alpha RNA expression | At baseline and in weeks 6, 7, and 13
  IL-6 and TNF-alpha measured from Peripheral blood mononuclear cell (PBMC)

SECONDARY OUTCOMES:
Doses of pancreatic enzyme replacement therapy | Only at baseline
  Measured in International Unit per day (IU/day)
Stool characteristics | At baseline and in weeks 6, 7, and 13
  The number and type of stools will be assessed using the Kings Stool Chart, a standardized tool that classifies stool consistency and form to evaluate digestive function alterations.
  * Number of bowel movements: A numerical field to record the daily count.
  * Type of bowel movements: A categorical field with options ranging from 1 to 7, based on the King's Stool Chart.
  * Variability in type: A binary field (0 = No, 1 = Yes) to indicate whether there is variation.
Symptoms of anxiety and depression | At baseline and in weeks 6, 7, and 13
  Measured using the Hospital Anxiety and Depression Scale (HADS), which consists of two subscales: HADS-Anxiety (HADSA) and HADS-Depression (HADSD)
  Interpretation of scores:
  * 0-7: Normal.
  * 8-10: Suggests the presence of mood disorders.
  * ≥11: Indicates a probable mood disorder.
Nutritional status | At baseline and in weeks 6, 7, and 13
  Evaluated using the Subjective Global Assessment (SGA) and Global Leadership Initiative on Malnutrition (GLIM) criteria, both validated tools for classifying malnutrition severity.
  Patients will be categorized as at risk of malnutrition or having moderate or severe malnutrition based on results.
Change in Phase angle (PhA) (Vectorial Bioimpedance Analysis (BIVA)) | At baseline and in weeks 6, 7, and 13
  Phase angle (PhA) measured in degrees (º)
Change in total body water (TBW) (Vectorial Bioimpedance Analysis (BIVA)) | At baseline and in weeks 6, 7, and 13
  Total body water (TBW) measured in liters (l)
Change in extracellular water (ECW) (Vectorial Bioimpedance Analysis (BIVA)) | At baseline and in weeks 6, 7, and 13
  Extracellular water (ECW) measured in liters (l)
Change in intracellular water (ICW) (Vectorial Bioimpedance Analysis (BIVA)) | At baseline and in weeks 6, 7, and 13
  Intracellular water (ICW) measured in liters (l)
Change in Fat-free mass (FFM) (Vectorial Bioimpedance Analysis (BIVA)) | At baseline and in weeks 6, 7, and 13
  Fat-free mass (FFM) measured in kilograms (kg) and percentage (%)
Change in Fat mass (FM) (Vectorial Bioimpedance Analysis (BIVA)) | At baseline and in weeks 6, 7, and 13
  Fat mass (FM) measured in kilograms (kg) and percentage (%)
Change in Body cell mass (BCM) (Vectorial Bioimpedance Analysis (BIVA)) | At baseline and in weeks 6, 7, and 13
  Body cell mass (BCM) measured in kilograms (kg)
Change in appendicular skeletal muscle mass (ASMM) (Vectorial Bioimpedance Analysis (BIVA)) | At baseline and in weeks 6, 7, and 13
  Appendicular skeletal muscle mass (ASMM) measured in kilograms (kg)
Change in skeletal muscle index (SMI) (Vectorial Bioimpedance Analysis (BIVA)) | At baseline and in weeks 6, 7, and 13
  Skeletal muscle index (SMI) measured in kilogram per square meter (kg/m²)
Change in hydration (Vectorial Bioimpedance Analysis (BIVA)) | At baseline and in weeks 6, 7, and 13
  Hydration measured in percentage (%)
Change in resistance (Vectorial Bioimpedance Analysis (BIVA)) | At baseline and in weeks 6, 7, and 13
  Resistance measured in ohms (Ω)
Change in reactance (Vectorial Bioimpedance Analysis (BIVA)) | At baseline and in weeks 6, 7, and 13
  Reactance measured in ohms (Ω)
Handgrip dynamometry | At baseline and in weeks 6, 7, and 13
  * Device: Jamar hydraulic dynamometer
  * Measurement:
  Mean and maximum grip strength (kg) from three measurements Used to assess sarcopenia
Timed Up and Go (TUG) Test | At baseline and in weeks 6, 7, and 13
  * Measures mobility and physical function
  * Procedure: Time (seconds) taken for the patient to:
    1. Rise from a chair
    2. Walk a short distance
    3. Return to the chair
Change in total fat (Abdominal Ultrasound) | At baseline and in weeks 6, 7, and 13
  Total fat measured in centimeters (cm)
Change in superficial fat (Abdominal Ultrasound) | At baseline and in weeks 6, 7, and 13
  Superficial fat measured in centimeters (cm)
Change in preperitoneal fat (Abdominal Ultrasound) | At baseline and in weeks 6, 7, and 13
  Preperitoneal fat measured in centimeters (cm)
Change in muscle Ultrasound - Area | At baseline and in weeks 6, 7, and 13
  Area measured in square centimeters (cm²)
Change in muscle Ultrasound - Circumference | At baseline and in weeks 6, 7, and 13
  Circumference measured in centimeters (cm)
Change in muscle Ultrasound - X-axis and Y-axis | At baseline and in weeks 6, 7, and 13
  X-axis and Y-axis measured in centimeters (cm)
Change in muscle Ultrasound - Adipose tissue of the rectus femoris of the quadriceps | At baseline and in weeks 6, 7, and 13
  Adipose tissue of the rectus femoris of the quadriceps measured in centimeters (cm)
Change in Glucose | At baseline and in weeks 6, 7, and 13
  glucose measured in mg/dl
Change in Cholesterol | At baseline and in weeks 6, 7, and 13
  Cholesterol measured in mg/dl
Change in Triglycerides | At baseline and in weeks 6, 7, and 13
  Triglycerides measured in mg/dl
Change in Uric acid | At baseline and in weeks 6, 7, and 13
  Uric acid measured in mg/dl
Change in AST | At baseline and in weeks 6, 7, and 13
  AST measured in units per litre (U/L)
Change in ALT | At baseline and in weeks 6, 7, and 13
  ALT measured in units per litre (U/L)
Change in GGT | At baseline and in weeks 6, 7, and 13
  GGT measured in units per litre (U/L)
Change in ALP | At baseline and in weeks 6, 7, and 13
  ALP measured in units per litre (U/L)
Change in insulin | At baseline and in weeks 6, 7, and 13
  Insulin measured in units per mililitre (U/mL)
Change in albumin | At baseline and in weeks 6, 7, and 13
  Albumin measured in grams per liter (g/l)
Change in C-reactive protein (CRP) | At baseline and in weeks 6, 7, and 13
  C-reactive protein (CRP) measured in milligrams per liter (mg/L)
Change in Intestinal fatty acid-binding protein (I-FABP) | At baseline and in weeks 6, 7, and 13
  Intestinal fatty acid-binding protein (I-FABP) measured in picograms per milliliter (pg/mL)
Change in zonulin | At baseline and in weeks 6, 7, and 13
  Zonulin measured in micrograms per milliliter (μg/mL)
Change in musclin | At baseline and in weeks 6, 7, and 13
  Musclin measured in nanograms per milliliter (ng/mL)
Change in galectin-3 | At baseline and in weeks 6, 7, and 13
  Galectin-3 measured in nanograms per milliliter (ng/mL)
Change in myostatin | At baseline and in weeks 6, 7, and 13
  Myostatin measured in nanograms per milliliter (ng/mL)
Change in Total antioxidant capacity (TAC) | At baseline and in weeks 6, 7, and 13
  Total antioxidant capacity (TAC) measured in nanomoles per microliter (nmol/μL)
Change in Glutathione peroxidase (GSH-Px) | At baseline and in weeks 6, 7, and 13
  Glutathione peroxidase (GSH-Px) measured in milliunits per milliliter (mU/mL)
Change in Superoxide dismutase (SOD) | At baseline and in weeks 6, 7, and 13
  Superoxide dismutase (SOD) measured in inhibition rate %
Change in GLP-1 | At baseline and in weeks 6, 7, and 13
  GLP-1 measured in picograms per milliliter (pg/mL)
Change in GIP | At baseline and in weeks 6, 7, and 13
  GIP measured in picograms per milliliter (pg/mL)
Change in PYY | At baseline and in weeks 6, 7, and 13
  PYY measured in picograms per milliliter (pg/mL)
Change in IFN-gamma | At baseline and in weeks 6, 7, and 13
  IFN-gamma measured in picograms per milliliter (pg/mL)
Change in IL-2 | At baseline and in weeks 6, 7, and 13
  IL-2 measured in picograms per milliliter (pg/mL)
Change in IL-4 | At baseline and in weeks 6, 7, and 13
  IL-4 measured in picograms per milliliter (pg/mL)
Change in IL-6 | At baseline and in weeks 6, 7, and 13
  IL-6 measured in picograms per milliliter (pg/mL)
Change in IL-10 | At baseline and in weeks 6, 7, and 13
  IL-10 measured in picograms per milliliter (pg/mL)
Change in IL-12p70 | At baseline and in weeks 6, 7, and 13
  IL-12p70 measured in picograms per milliliter (pg/mL)
Change in IL-17A | At baseline and in weeks 6, 7, and 13
  IL-17A measured in picograms per milliliter (pg/mL)
Change in TNF-alpha | At baseline and in weeks 6, 7, and 13
  TNF-alpha measured in picograms per milliliter (pg/mL)
Change in stool calprotectin | At baseline and in weeks 6, 7, and 13
  Calprotectin measured in micrograms per gram (µg/g)

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Olveira Fuster, MD, PhD, Principal Investigator — Hospital Regional Universitario de Málaga, FIMABIS
Locations (1):
- Hospital Regional Universitario de Málaga, Málaga, Málaga, Spain

IPD SHARING:
Plan to Share IPD: No
It is not necessary to reach the objectives of the project